CLINICAL TRIAL: NCT03610672
Title: Preventing Injection: An mHealth Intervention That Leverages Social Networks to Prevent Progression to Injection Among Young Opioid Users
Brief Title: Mobile Intervention for Young Opioid Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R34DA043957 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The current study is a two-armed, open randomized clinical trial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OD prevention/response training (Active Comparator): Immediately following the baseline assessment, trained research staff will conduct a brief (20 min.) OD training with each participant. Participants will be asked to view the NYC Department of Health and Mental Hygiene's 13-minute OD prevention and response training video (available online free-of-charge). Following the video, research staff will review key information, answer any questions participants may have, demonstrate assembly of the intranasal naloxone atomizer and ensure participants are able to execute this assembly procedure. A prescription for naloxone, as well as a standard naloxone kit containing two doses of the medication and atomizers for intranasal administration, will be given to participants, along with printed literature reviewing key training information.
  Interventions: Behavioral: OD prevention/response training
- OD training + mobile PI intervention (Experimental): Participants will complete the same baseline assessment and OD training (plus naloxone) as those in the first condition. Participants also will receive mobile phones pre-loaded with the PI App and will be sent daily prompts. As part of the PI App, participants will be asked to share information about avoiding problems associated with opioid use with peers in their social network, and to encourage their peers to download the PI App for their own use.
  Interventions: Behavioral: OD prevention/response training + PI mobile application

INTERVENTIONS:
Behavioral: OD prevention/response training — Participants will view a 13-minute OD prevention and response training video (available online free-of-charge). This video covers NY State's recommended curriculum for Overdose Prevention: how to prevent, identify, and respond to an OD, including information on the factors that could heighten risk for overdose (mixing drugs, changes in tolerance and drug purity, and using alone), how to respond to an overdose (rescue breathing, calling 911), and specific instructions on how and when to administer naloxone to someone who is overdosing. After the video, research staff will review key information, answer any questions participants may have, demonstrate assembly of the intranasal naloxone atomizer and ensure participants are able to assemble it. A prescription for naloxone, as well as a standard naloxone kit containing two doses of the medication and atomizers for intranasal administration, will be given to participants, along with printed literature reviewing key training information.
  Arms: OD prevention/response training
Behavioral: OD prevention/response training + PI mobile application — Participants will receive the same OD intervention as those in the first arm, as well as receiving mobile phones pre-loaded with the PI App. This intervention includes daily prompts plus key components of evidence-based cognitive behavioral interventions, including Functional Analysis of Drug Use, Self-Management, and Social/Recreational Counseling and additional content on Distress Tolerance, the relationship between Peer Networks and Drug Use, and pertinent resources.
  Arms: OD training + mobile PI intervention

SUMMARY:
Opioid use disorders (OUD) are the second most common type of drug use disorder in the US, with nearly 2 million Americans with prescription opioid- (PO) and ~570,000 with heroin-related OUD. The escalation in OUD during the past two decades has been most pronounced among youth, many of whom demonstrate a rapid transition from nonmedical PO use (16-17 y/o), to heroin (19-20 y/o), with most progressing to injection drug use (IDU), within a year of starting heroin use (20-21 y/o). Progression to IDU is characterized by uniquely high levels of risk for youth, including higher rates of overdose (OD) and HIV and HCV incidence, compared to older peers. Addiction severity, psychosocial functioning, and social networks are robust predictors of transitioning to IDU; however there is virtually no research on how to prevent or halt this transition to IDU. Given the paucity of interventions targeting this large and vulnerable group of youth, we propose to adapt and evaluate an innovative, engaging mHealth intervention to prevent young opioid users (18-29) from transitioning to IDU. Aim 1: During months 1-12, we will adapt our existing mobile intervention for OUD that includes daily text messages plus key components of evidence-based CBT interventions, including Functional Analysis of Drug Use, Self-Management, and Social / Recreational Counseling. New components specific to youth will focus on the role of peers on opioid use and IDU, and OD prevention / response training. Our iterative development process will include focus groups with opioid-using youth (n=24), interviews with important stakeholders (e.g., youth treatment providers; n=6), and feedback and usability data from opioid-using youth (n=30). Aim 2: During months 13-31, we will conduct a small randomized, controlled trial of the tailored mHealth intervention with young opioid users who have not transitioned to regular injection (n=64) and compare (1) assessment plus in-person OD prevention / response training (including naloxone) versus (2) assessment plus in-person OD prevention / response training (including naloxone) plus our mHealth intervention. Feasibility and acceptability will be assessed via participant feedback, retention, and usage data. Diffusion will be defined as the number of participants' peers who download the intervention app for their own use. Preliminary effectiveness will be measured via reductions in opioid use (TLFB, urine / hair toxicology) and self-reported injection status at 4, 8, and 12 weeks, and 3 and 6 month follow-up. Secondary outcomes include HIV/HCV risk behavior, OD, opioid-related problems (e.g., withdrawal episodes), and social network IDU-related norms and behaviors. If results are promising, this novel intervention will be expanded for examination in a large-scale efficacy / effectiveness trial.

DETAILED DESCRIPTION:
Opioid use disorders (OUD) are the second most common type of drug use disorder in the US, with nearly 2 million reporting prescription opioid (PO) use and ~570,000 reporting heroin use consistent with an OUD. Further, drug overdose (OD) has become the leading cause of accidental death in the US, with opioid-involved OD driving this epidemic. The recent escalation in OUD has been most pronounced among youth, with nearly 1/3 of youth reporting PO misuse by age 21, and studies have documented the trajectory from PO misuse to injection drug use (IDU) in youth. An ongoing study conducted by the current investigators documented an alarming trajectory, wherein these youth progress from nonmedical PO use in adolescence (first PO use M=16.7 y/o), to oral / intranasal heroin use in young adulthood (M=19.1 y/o), with 64% progressing to injection drug use (IDU), within a year of heroin initiation (first injection M=20.1 y/o. This progression to IDU is characterized by uniquely high levels of risk for youth, including higher rates of injection risk behaviors and OD, and higher incidence of HIV and HCV within the first few years of transitioning to injection, compared to older peers. Thus, young opioid users are at uniquely high risk for a number of negative outcomes during the critical period of transitioning to injection. This rapid progression from PO use to IDU and the extreme risk associated with new injection status among youth indicate that there is a brief, but critical, period during which we may intervene to prevent progression to injection and its associated risk behaviors and negative health outcomes. Several robust predictors have been found for progression to IDU, including psychosocial factors (i.e., homelessness, physical abuse), OUD severity (i.e., dependence severity, polydrug use), and IDU norms and behaviors within one's social network. While there is some understanding of the mechanisms that promote IDU, there is virtually no research on strategies to prevent this transition. Only one intervention has been examined targeting intranasal heroin users in an attempt to prevent progression to IDU. This "sniffers" intervention found potent effects; half as many intervention participants progressed to injection (33% vs. 16%), compared to the control condition (who received HIV/AIDS education), indicating that direct intervention with opioid users may be an effective way to prevent progression to IDU and its associated harms. It is unclear why so few interventions have targeted this population, although young opioid users face a number of unique barriers, including social, economic, and motivational, that may prevent them from seeking and receiving treatment. Given the paucity of interventions available to the large and vulnerable group of opioid-using young adults, there is an urgent need to develop and evaluate innovative, engaging approaches to prevent young opioid users from transitioning to IDU.

The current application is being submitted in response to PA 16-073, "Behavioral and Integrative Treatment Development Program." The proposed project is a Stage Ib study that will adapt a mobile, evidence-based psychosocial intervention for opioid dependence (Check-In App) to prevent progression to injection in young opioid users (18-29 y/o) who have not progressed to regular injection.

Aim 1: During months 1-12, we will adapt the Check-In App to target reducing opioid use and preventing progression to injection among young oral / intranasal opioid users. We will tailor our existing mHealth intervention (including daily text messages plus key components of evidence-based cognitive behavioral interventions, Functional Analysis of Drug Use, Self-Management, and Social / Recreational Counseling), for young opioid users. New components specific to youth will focus on the role of peers in opioid use / IDU, and OD prevention / response training including use of naloxone. Our iterative development process will include focus groups with opioid-using youth (n=24), interviews with important stakeholders (e.g., youth treatment providers; n=6), and feedback and usability data from opioid-using youth (n=30).

Aim 2: During months 13-31, we will conduct a small randomized, controlled trial of the newly tailored mHealth intervention with young opioid users (18-29 y/o) who have not transitioned to regular injection (n=64) and compare (1) assessment plus in-person OD prevention / response training (including naloxone) versus (2) assessment plus in-person OD prevention / response training (including naloxone) plus the Preventing Injection Application. We will evaluate the intervention's feasibility, acceptability, diffusion, and preliminary effectiveness. Feasibility and acceptability will be assessed via participant feedback, retention, and app usage data. Diffusion will be defined as the number of participants' peers who download the intervention app for their own use. Preliminary effectiveness will be measured via reductions in opioid use (TLFB, urine and hair toxicology) and self-reported injection status at 4, 8, and 12 weeks, and 3 and 6 month follow-up. Secondary outcomes include HIV/HCV risk behavior, OD episodes, opioid-related problems (e.g., withdrawal episodes), and social network IDU-related norms and behaviors.

If results are promising, this intervention will be evaluated in a large-scale efficacy / effectiveness trial. This intervention may have tremendous impact on improving access, acceptability, and potency of opioid use interventions for youth, given the extremely widespread use of mobile apps among young adults (98% of 18-29 y/o own mobile phones and spend ~3 hr/day using mobile apps).

ELIGIBILITY:
Inclusion Criteria:

* Current opioid use, defined as having used heroin and/or POs 12 or more times in the past 30 days (self-report verified by urine toxicology)
* Aged 18-29 years, verified by photo ID
* Able to understand and speak English
* Willing and available to participate in the assigned intervention.

Exclusion Criteria:

* Individuals are excluded if they report regular injection drug use (defined as injection 3 or more times/week in the past 30 days) for a period of more than 24 months

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-11-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in opioid use | Change from baseline to 12 weeks
  Participant opioid use will be assessed via self-reported Timeline Followback, urine toxicology, and hair toxicology
Change in self-reported injection status via Timeline Followback | Change from baseline to 12 weeks
  Self-reports of frequency and duration of injection drug use

SECONDARY OUTCOMES:
Change in HIV/HCV risk behavior | Change from baseline to 12 weeks
  self-reported HIV/HCV risk behavior (combined injection and sexual risk behavior)
OD | 12 weeks
  frequency and severity of self-reported overdose (OD) episodes
Peer IDU norms | Change from baseline to 12 weeks
  Self-reported perceptions of peer injection drug use-related norms

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Acosta, Principal Investigator — NIDA/NIH
Locations (1):
- National Development and Research Institutes, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No